CLINICAL TRIAL: NCT00003890
Title: A Phase I Study of MG98 Given as a 2 Hour Twice Weekly IV Infusion in Patients With Advanced Cancer
Brief Title: MG98 in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I125; CAN-NCIC-IND125 (Other: PDQ); METHYL-MG98-002 (Other: Methylgene Inc.); CDR0000067059 (Other: PDQ)
Record Dates: First submitted 2000-06-02; First posted 2003-08-20 (Estimated); Last update posted 2020-04-06 (Actual); Status verified 2020-04

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: MG 98

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of MG98 in treating patients who have advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of MG98 in patients with advanced solid tumors.
* Assess the safety, toxicity, and pharmacokinetics of this treatment regimen in this patient population.
* Evaluate the effectiveness of this treatment regimen in these patients.

OUTLINE: This is a dose escalation, multicenter study.

Patients receive MG98 IV over 2 hours twice weekly for 3 weeks. Courses are repeated every 4 weeks. Treatment continues in the absence of disease progression or unacceptable toxicity.

The dose of MG98 is escalated in cohorts of 1-6 patients until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose limiting toxicity.

Patients are followed at week 4, then at least every 3 months until relapse of disease.

PROJECTED ACCRUAL: Approximately 20 patients will be accrued for this study within 10-12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically proven advanced solid tumor unresponsive to existing therapy or for which no curative therapy exists
* Evidence of disease in addition to tumor marker elevation
* CNS metastases allowed, if adequately treated and symptoms controlled for greater than 4 months

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* At least 12 weeks

Hematopoietic:

* Absolute granulocyte count at least 1,500/mm3
* Platelet count at least 100,000/mm3
* PTT normal

Hepatic:

* Bilirubin no greater than 1.25 times upper limit of normal (ULN)
* SGOT or SGPT no greater than 3 times ULN (4 times ULN for liver metastases)

Renal:

* Creatinine no greater than 1.25 times ULN
* Proteinuria less than 2+ (no greater than 500 mg in a 24 hour urinalysis)

Other:

* No active infection
* No other serious systemic disease
* No known hypersensitivity to oligodeoxynucleotides
* Adequate venous access
* No known condition (e.g., psychological, geographical) that would prevent compliance
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after the study

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent colony stimulating factors unless evidence of neutropenic infection

Chemotherapy:

* No more than 3 prior chemotherapy regimens
* At least 3 weeks since prior chemotherapy (6 weeks for nitrosoureas and mitomycin) and recovered
* At least 1 year since prior high dose chemotherapy with bone marrow or stem cell support
* No concurrent chemotherapy

Endocrine therapy:

* Prior hormonal therapy allowed
* No concurrent hormonal therapy

Radiotherapy:

* At least 4 weeks since prior radiotherapy and recovered
* Concurrent palliative radiotherapy allowed

Surgery:

* At least 2 weeks since prior major surgery

Other:

* At least 3 weeks since prior investigational drug therapy
* No other concurrent investigational drug or anticancer therapy
* No concurrent coumadin or heparin therapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 1999-02-22 (Actual); Primary Completion 2001-09-27 (Actual); Study Completion 2008-09-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ross C. Donehower, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (2):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States
- Ottawa Regional Cancer Centre, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Stewart DJ, Donehower RC, Eisenhauer EA, Wainman N, Shah AK, Bonfils C, MacLeod AR, Besterman JM, Reid GK. A phase I pharmacokinetic and pharmacodynamic study of the DNA methyltransferase 1 inhibitor MG98 administered twice weekly. Ann Oncol. 2003 May;14(5):766-74. doi: 10.1093/annonc/mdg216. PMID 12702532